CLINICAL TRIAL: NCT00777491
Title: A Phase II Randomized Study For Patients With Muscle-Invasive Bladder Cancer Evaluating Transurethral Surgery And Concomitant Chemoradiation By Either BID Irradiation Plus 5-Fluorouracil And Cisplatin Or QD Irradiation Plus Gemcitabine Followed By Selective Bladder Preservation And Gemcitabine/Cisplatin Adjuvant Chemotherapy
Brief Title: Chemotherapy and Radiation Therapy in Treating Patients With Stage II or Stage III Bladder Cancer That Was Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0712; CDR0000616858
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; stage III bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Fluorouracil; Gemcitabine; Cisplatin; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-FU and Cisplatin + BID Irradiation (Experimental): Within 8 weeks following pre-study transurethral resection (TUR) patients receive 2.5 weeks of induction chemoradiotherapy (induction 5-fluorouracil, induction cisplatin, induction BID radiation therapy). Consolidation chemoradiotherapy begins 7-14 days following post-induction chemoradiotherapy endoscopic response evaluation. Patients achieving a complete response receive 1.5 weeks of consolidation chemoradiotherapy (consolidation 5-fluorouracil, consolidation cisplatin, consolidation BID radiation therapy). Patients without a complete response undergo radical cystectomy. Outpatient adjuvant chemotherapy (adjuvant gemcitabine, adjuvant cisplatin) begins 4-5 weeks following the post-consolidation endoscopic evaluation or 8-12 weeks following radical cystectomy, and continues for 12 weeks.
  Interventions: Drug: induction cisplatin; Drug: induction 5-fluorouracil; Radiation: Induction BID radiation therapy; Radiation: Consolidation BID radiation therapy; Drug: consolidation 5-fluorouracil; Drug: consolidation cisplatin; Procedure: radical cystectomy; Procedure: Post-Induction Chemoradiotherapy Endoscopic Response Evaluation; Drug: adjuvant gemcitabine; Drug: adjuvant cisplatin
- Gemcitabine + QD Irradiation (Experimental): Within 8 weeks following pre-study transurethral resection (TUR) patients receive 2.5 weeks of induction chemoradiotherapy (induction gemcitabine and induction QD radiation therapy). Consolidation chemoradiotherapy begins 7-14 days following post-induction chemoradiotherapy endoscopic response evaluation. Patients achieving a complete response receive 1.5 weeks of consolidation chemoradiotherapy (consolidation gemcitabine and consolidation QD radiation therapy). Patients without a complete response undergo radical cystectomy. Outpatient adjuvant chemotherapy (adjuvant gemcitabine and adjuvant cisplatin) begins 4-5 weeks following the post-consolidation endoscopic evaluation or 8-12 weeks following radical cystectomy, and continues for 12 weeks.
  Interventions: Drug: induction gemcitabine; Radiation: Induction QD radiation therapy; Radiation: Consolidation QD radiation therapy; Drug: consolidation gemcitabine; Procedure: radical cystectomy; Procedure: Post-Induction Chemoradiotherapy Endoscopic Response Evaluation; Drug: adjuvant gemcitabine; Drug: adjuvant cisplatin

INTERVENTIONS:
Drug: induction cisplatin — 15 mg/m^2 administered as a 60-minute infusion on days 1,2,3,8,9,10,15,16,17.
  Arms: 5-FU and Cisplatin + BID Irradiation
Drug: induction 5-fluorouracil — 400mg/m^2 administered as a 24-hour infusion on days 1,2,3, and 15,16,17.
  Other Names: fluorouracil; 5-FU
  Arms: 5-FU and Cisplatin + BID Irradiation
Drug: induction gemcitabine — 27 mg/m^2 administered as a 30-minute infusion on days 1, 4, 8, 11, 15, 18, 22, 25.
  Other Names: gemcitabine hydrochloride
  Arms: Gemcitabine + QD Irradiation
Radiation: Induction BID radiation therapy — Twice daily (BID) on days 1-5,8-12,15-17. The first daily treatment consists of 1.6 Gy delivered to the pelvis. The second fraction consists of 1.5 Gy to the bladder for the first 5 treatment days. Then, 1.5 Gy is delivered to bladder tumor volume as the second treatment for the remaining 8 treatment days. The bladder tumor volume receives a total of 40.3 Gy.
  Arms: 5-FU and Cisplatin + BID Irradiation
Radiation: Induction QD radiation therapy — Once daily (QD) on days (1-5,8-12,15-19,22-26). For the first 10 treatment days, 2 Gy is delivered to the pelvis. Then, 2 Gy is delivered to the bladder for the next 4 treatment days, followed by 2 Gy to the bladder tumor volume for the remaining 6 treatment days. The bladder tumor volume receives a total of 40 Gy.
  Arms: Gemcitabine + QD Irradiation
Radiation: Consolidation BID radiation therapy — Twice daily (BID) for 8 days on days 1,2,3,4,5,8,9,10 of consolidation. 1.5 Gy per fraction for a total of 24 Gy delivered to the pelvis.
  Arms: 5-FU and Cisplatin + BID Irradiation
Radiation: Consolidation QD radiation therapy — Once daily (QD) pelvic radiation therapy for 12 days on days 1-5,8-12,15-16 of consolidation. 2 Gy per fraction for a total of 24 Gy delivered to the pelvis.
  Arms: Gemcitabine + QD Irradiation
Drug: consolidation gemcitabine — 27 mg/m^2 administered as a 30-minute infusion on days 1, 4, 8, 11, 15 of consolidation.
  Other Names: gemcitabine hydrochloride
  Arms: Gemcitabine + QD Irradiation
Drug: consolidation 5-fluorouracil — 400 mg/m^2 administered as a 24-hour infusion on days 1, 2, 3 and 8, 9, 10 of consolidation.
  Other Names: fluorouracil; 5-FU
  Arms: 5-FU and Cisplatin + BID Irradiation
Drug: consolidation cisplatin — 15 mg/m^2 administered as a sixty-minute infusion on days 1, 2, 8, 9 of consolidation.
  Other Names: cisplatin
  Arms: 5-FU and Cisplatin + BID Irradiation
Procedure: radical cystectomy — Operable patients who have a pT1 or worse tumor response on re-evaluation following initial transurethral resection and induction chemoradiotherapy will have a radical cystectomy 3-8 weeks following the post-induction response evaluation.
Procedure: Post-Induction Chemoradiotherapy Endoscopic Response Evaluation — Urine cytology, cystoscopy, tumor site transurethral biopsy, and bimanual examination after biopsy.
  Other Names: TUR
Drug: adjuvant gemcitabine — 1000 mg/m^2 administered intravenously over 30-60 minutes (preferably 30 minutes) on days 1 and 8 of each 21-day cycle for four cycles.
  Other Names: gemcitabine hydrochloride
Drug: adjuvant cisplatin — 70 mg/m^2 administered as a sixty-minute infusion on day 1 of each 21-day cycle for four cycles.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, cisplatin, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying two different chemotherapy and radiation therapy regimens to see how they work in treating patients with stage II or stage III bladder cancer that was removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the rate of distant metastasis at 3 years in patients who have undergone transurethral resection of the bladder tumor for stage II or III muscle-invasive bladder cancer treated with chemoradiotherapy comprising fluorouracil, cisplatin, and radiotherapy vs gemcitabine hydrochloride and radiotherapy followed by selective bladder preservation and adjuvant chemotherapy comprising gemcitabine hydrochloride and cisplatin.

Secondary

* To estimate the treatment completion rate in these patients.
* To estimate acute and late grade toxicities (≥ grade 3 genitourinary, gastrointestinal, and hematologic toxicities) of these regimens in these patients.
* To estimate the efficacy of these regimens, in terms of achieving complete response of the primary tumor, in these patients.
* To estimate the efficacy of these regimens, in terms of preserving the native, tumor-free bladder 5 years after completion of therapy, in these patients.
* To estimate the value of tumor histopathologic, molecular genetic, DNA content, metabolomic, and proteomic parameters as possible significant prognostic factors for initial tumor response and recurrence-free survival.
* To analyze for American Urological Association (AUA) Symptom scores at baseline and at 3 years from patients on both arms.
* To find potentially predictive biomarkers for cystectomy-free survival.
* To find potentially predictive biomarkers for acute and late toxicities.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor stage (T2 vs T3-4a). Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically (histologically or cytologically) proven diagnosis of primary carcinoma of the bladder (transitional cell cancer) within 8 weeks of registration. Operable patients whose tumors are primary carcinomas of the bladder and exhibit histologic evidence of muscularis propria invasion and are American Joint Committee on Cancer (AJCC) clinical stages T2-T4a, Nx or N0, M0 (Appendix IV) without hydronephrosis; patients who have involvement of the prostatic urethra with transitional cell cancer (TCC) that was visibly completely resected and no evidence of stromal invasion of the prostate remain eligible. T2a, T2b, T3a, T3b -substages‖ are not usually able to be determined with clinical (TURBT) staging.
2. If radiologic evaluation of a lymph node is interpreted as "positive", this must be evaluated further either by lymphadenectomy or percutaneous needle biopsy. Patients with histologically or cytologically confirmed node metastases will not be eligible.
3. Patients must have an adequately functioning bladder after thorough evaluation by an urologist and have undergone as thorough a transurethral resection of the bladder tumor as is judged safely possible.
4. Patients must be considered able to tolerate systemic chemotherapy combined with pelvic radiation therapy, and a radical cystectomy by the joint agreement of the participating Urologist, Radiation Oncologist, and Medical Oncologist.
5. History and physical examination including weight, performance status, and body surface area within 8 weeks prior to study registration
6. Zubrod Performance Status ≤ 1
7. Age ≥ 18
8. Complete blood count (CBC)/differential obtained no more than 4 weeks prior to registration on study, with adequate bone marrow function defined as follows:

   * 8.1 White blood cell count (WBC) ≥ 4000/ml
   * 8.2 Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3;
   * 8.3 Platelets ≥ 100,000 cells/mm3;
   * 8.4 Hemoglobin (hgb) ≥ 10.0 mg/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10.0 g/dl is acceptable.);
9. Serum creatinine of 1.5 mg% or less; serum bilirubin of 2.0 mg% or less; creatinine clearance of 60 ml/min or greater no more than 4 weeks prior to registration; Note: Calculated creatinine clearance is permissible. If the creatinine clearance is > 60 ml/min, then a serum creatinine of up to 1.8 mg% is allowable at the discretion of the study chair;
10. Serum pregnancy test for female patients of childbearing potential, ≤ 72 hours prior to study entry; women of childbearing potential and male participants must practice adequate contraception.
11. Patient must be able to provide study-specific informed consent prior to study entry.

Exclusion criteria:

1. Evidence of tumor-related hydronephrosis
2. Evidence of distant metastases or histologically or cytologically proven lymph node metastases
3. Previous systemic chemotherapy (for any cancer) or pelvic radiation therapy
4. A prior or concurrent malignancy of any other site or histology unless the patient has been disease-free for ≥ 5 years except for non-melanoma skin cancer and/or stage T1a prostate cancer or carcinoma in situ of the uterine cervix
5. Patients judged not to be candidates for radical cystectomy; patients with pN+ or T4b disease are considered to have unresectable disease
6. Patients receiving any drugs that have potential nephrotoxicity or ototoxicity (such as an aminoglycoside)
7. Severe, active co-morbidity, defined as follows:

   * 7.1 Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
   * 7.2 Transmural myocardial infarction within the last 6 months;
   * 7.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
   * 7.4 Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
   * 7.5 Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
   * 7.6 Acquired Immune Deficiency Syndrome (AIDS) based upon current Center for Disease Control (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
8. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
9. Prior allergic reaction to the study drug(s) involved in this protocol

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-12; Primary Completion 2018-02-18 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J. Coen, MD, Principal Investigator — GenesisCare USA; Philip J. Saylor, MD, Study Chair — Massachusetts General Hospital; Cheryl T. Lee, MD, Study Chair — University of Michigan Rogel Cancer Center; Chin-Lee Wu, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (11):
- United States (10):
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
- McGill Cancer Centre at McGill University, Montreal, Quebec, Canada

REFERENCES:
- [Result] Choudhury A, Swindell R, Logue JP, Elliott PA, Livsey JE, Wise M, Symonds P, Wylie JP, Ramani V, Sangar V, Lyons J, Bottomley I, McCaul D, Clarke NW, Kiltie AE, Cowan RA. Phase II study of conformal hypofractionated radiotherapy with concurrent gemcitabine in muscle-invasive bladder cancer. J Clin Oncol. 2011 Feb 20;29(6):733-8. doi: 10.1200/JCO.2010.31.5721. Epub 2011 Jan 4. PMID 21205754

RESULTS

PARTICIPANT FLOW:
Groups:
- 5-FU and Cisplatin + BID Irradiation: Within 8 weeks following pre-study transurethral resection (TUR) patients receive 2.5 weeks of induction chemoradiotherapy (induction 5-fluorouracil, induction cisplatin, induction BID [twice daily] radiation therapy). Consolidation chemoradiotherapy begins 7-14 days following post-induction chemoradiotherapy endoscopic response evaluation. Patients achieving a complete response receive 1.5 weeks of consolidation chemoradiotherapy (consolidation 5-fluorouracil, consolidation cisplatin, consolidation BID radiation therapy). Patients without a complete response undergo radical cystectomy. Outpatient adjuvant chemotherapy (adjuvant gemcitabine, adjuvant cisplatin) begins 4-5 weeks following the post-consolidation endoscopic evaluation or 8-12 weeks following radical cystectomy, and continues for 12 weeks.
- Gemcitabine + QD Irradiation: Within 8 weeks following pre-study transurethral resection (TUR) patients receive 2.5 weeks of induction chemoradiotherapy (induction gemcitabine and induction QD [once a day] radiation therapy). Consolidation chemoradiotherapy begins 7-14 days following post-induction chemoradiotherapy endoscopic response evaluation. Patients achieving a complete response receive 1.5 weeks of consolidation chemoradiotherapy (consolidation gemcitabine and consolidation QD radiation therapy). Patients without a complete response undergo radical cystectomy. Outpatient adjuvant chemotherapy (adjuvant gemcitabine and adjuvant cisplatin) begins 4-5 weeks following the post-consolidation endoscopic evaluation or 8-12 weeks following radical cystectomy, and continues for 12 weeks.
Period: Overall Study
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation
Started | 35 | 35
Eligible | 33 | 33
Has 3-year Efficacy Data (Eligible and has 3-year distant metastasis status) | 27 | 25
Started Induction Therapy (Eligible and started induction therapy) | 33 | 33
Started Consolidation Therapy (Eligible and started consolidation therapy) | 29 | 25
Started Adjuvant Therapy (Eligible and started adjuvant therapy) | 32 | 31
Has Adverse Event Data (Treatment) (Eligible and has adverse event data during treatment) | 33 | 33
Has Adverse Event Data (Late) (Eligible and has adverse event data between end of treatment to 180 days after end of treatment) | 32 | 31
Has 3 Year AUASI Data (Eligible and has baseline and 3-year American Urological Association Symptom Index (AUASI) scores) | 6 | 6
Completed (Subjects contributing any data to analysis are considered to have completed the study) | 33 | 33
Not Completed | 2 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Did not receive any protocol treatment | 2 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Customized [Count of Participants; unit: Participants]
  <= 49 years | 2 | 0 | 2
  50-59 years | 5 | 4 | 9
  60-69 years | 13 | 20 | 33
  >= 70 years | 13 | 9 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 32 | 33 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 30 | 29 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Zubrod Performance Status [Count of Participants; unit: Participants] — Measure Description: 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 29 | 32 | 61
    1 | 4 | 1 | 5
T Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    cT2 | 32 | 32 | 64
    cT3-T4a | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Without Distant Metastases by Three Years
Description: Distant metastasis occurrence is defined as the first appearance of disease (with radiographic evidence) in a non-regional lymph node, solid organ or bone.
Time Frame: From randomization to three years
Population: Eligible patients with 3-year data
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation
Number analyzed (Participants) | 27 | 25
percentage of participants | 77.8 [64.3 to NA] — One-sided confidence interval | 84.0 [70.5 to NA] — One-sided confidence interval
Statistical Analysis 1: Comparison: 5-FU and Cisplatin + BID Irradiation vs Gemcitabine + QD Irradiation; The confidence interval of the rate was calculated by Clopper-Pearson's exact binomial confidence intervals methods with one-sided type I error of 0.1. The study required 32 analyzable patients in each arm, which would warrant a 10% chance of observing a percentage of patients without distant metastasis by 3 years of less than 75% if the true rate was 86%. With the actual number of evaluable patients, the study instead warrants a 13-14% chance; Test type: Other — There was no formal comparison of the two treatment arms; If the percentage of patients without distant metastasis by 3 years for either arm was greater than or equal to 75%, then it would be strongly considered as a potential arm in a subsequent phase III study, assuming treatment delivery and adverse events (AEs) were acceptable. If both arms met the criteria, then the treatment arm with less toxicity would be chosen

2. Secondary Outcome: Percentage of Patients Who Completed Treatment Per Protocol
Description: Treatment administration data was centrally reviewed to determine if patients completed each treatment component per protocol.
Time Frame: After each treatment component (induction, consolidation, adjuvant). Timing varies bases on arm, tumor response at multiple time points, and allowed time ranges.
Population: Eligible patients who started each treatment component (induction, consolidation, adjuvant)
Measure: Count of Participants; unit: Participants
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation
Number analyzed (Participants) | 33 | 33
Participants
  Induction Therapy | 32 | 31
  Consolidation Therapy: number analyzed (Participants) | 29 | 25
  Consolidation Therapy | 27 | 23
  Adjuvant Therapy: number analyzed (Participants) | 32 | 31
  Adjuvant Therapy | 18 | 17

3. Secondary Outcome: Percentage of Patients With Grade 3 or Higher Genitourinary, Gastrointestinal, or Hematologic Adverse Events
Description: Highest grade adverse event (AE) per subject was counted. Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. All adverse events are counted, regardless of reported relationship to protocol treatment.
Time Frame: From start of treatment to 180 days after the end of treatment. Treatment could last up to 40 weeks depending on arm, tumor response, and allowed time ranges.
Population: Eligible patients with adverse event data for corresponding time period
Measure: Count of Participants; unit: Participants
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation
Number analyzed (Participants) | 33 | 33
Participants
  During Treatment | 19 | 18
  Between End of Treatment and 180 days after: number analyzed (Participants) | 32 | 31
  Between End of Treatment and 180 days after | 8 | 5

4. Secondary Outcome: Number of Patients Experiencing Complete Response of the Primary Tumor After Induction Therapy
Description: Patients will be considered as having a clinical complete response when all biopsies are negative at the site(s) of the pretreatment tumor(s).
Time Frame: 3-4 weeks following induction therapy (approximately maximum 8 weeks from start of treatment depending on treatment arm and allowed time windows)
Population: Eligible patients who started induction therapy
Measure: Count of Participants; unit: Participants
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation
Number analyzed (Participants) | 33 | 33
Participants | 29 | 25
Statistical Analysis 1: Comparison: 5-FU and Cisplatin + BID Irradiation vs Gemcitabine + QD Irradiation; Test type: Superiority; p = 0.30, Regression, Logistic — Two-sided significance level of 0.05; Univariate analysis; Odds Ratio (OR) = 0.493, 95% CI 2-sided [0.129 to 1.881] — Reference arm = 5-FU and Cisplatin + BID Irradiation

5. Secondary Outcome: Number of Participants With Progression or Removal of Bladder Five Years After Therapy
Description: Progression is defined as an increase of 50% or more in the largest diameter of the endoscopically appreciable tumor in the tumor-site biopsy specimen, the development of new bladder tumors, or the development of metastatic disease.
Time Frame: From start of treatment to five years after the end of therapy. Treatment could last up to 40 weeks depending on arm, tumor response, and allowed time ranges.
Population: Eligible participants with five-year data
Measure: Count of Participants; unit: Participants
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation
Number analyzed (Participants) | 27 | 22
Participants | 4 | 5
Statistical Analysis 1: Comparison: 5-FU and Cisplatin + BID Irradiation vs Gemcitabine + QD Irradiation; Test type: Superiority; p = 0.75, Regression, Logistic — Two-sided significance level of 0.05; Univariable analysis; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.426 to 5.277] — Reference arm = 5-FU and Cisplatin + BID irradiation

6. Secondary Outcome: Change in American Urological Association Symptom Index (AUASI) Score at 3 Years
Description: The AUASI is a validated 7-item measure used to assess urinary symptoms. A higher score indicates more severe symptoms for the individual questions and overall total. Six questions ask about frequency of symptoms over the past month with possible responses: 0= Not at all; 1 = Less than 1 time in 5; 2 = less than half the time, 3 = About half the time, 4 = More than half the time, 5 = Almost always. An additional question asks the number of times one gets up to urinate after going to bed, with response indicating the exact number of times ranging from 0 to 5. The total score is the sum of the questions and ranges from 0 to 35. Change is calculated as 3-year score - baseline score such that a negative change indicates improvement.
Time Frame: Baseline and 3 years
Population: Eligible patients with baseline and 3-year scores
Measure: Median (Full Range); unit: units on a scale
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation
Number analyzed (Participants) | 6 | 6
units on a scale
  Sensation of Not Emptying Bladder | -0.50 [-4.00 to 0.00] | 0.0 [-3.00 to 3.00]
  Urinate Again < 2 Hours After Urinating | -2.50 [-5.00 to 2.00] | -1.0 [-4.00 to 4.00]
  Stopped and Started When Urinating | -1.00 [-5.00 to 1.00] | 0.00 [-1.00 to 2.00]
  Difficult to Postpone Urination | -3.00 [-5.00 to 0.00] | -0.50 [-3.00 to 4.00]
  Weak Urinary Stream | -0.50 [-5.00 to 0.00] | 0.00 [-2.00 to 5.00]
  Push or Strain to Begin Urination | -0.50 [-5.00 to 2.00] | 0.00 [-1.00 to 0.00]
  How Often Get Up at Night to Urinate | -3.50 [-4.00 to 4.00] | -1.50 [-2.00 to 4.00]
  AUA Total Symptom Score | -9.50 [-33.00 to 6.00] | -3.50 [-12.00 to 22.00]

7. Secondary Outcome: Determining Potentially Predictive Biomarkers for Acute and Late Toxicities
Time Frame: The protocol did not provide sufficient detail to meet National Cancer Institute requirements for release of specimens from the NRG tissue bank for the protocol-specified analysis, therefore no assays were performed and no data were collected for this out
Population: The protocol did not provide sufficient detail to meet National Cancer Institute requirements for release of specimens from our tissue bank for the protocol-specified analysis, therefore no assays were performed and no data were collected for this outcome measure. Specimen use will require federal approval and funding separate from this trial.
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Determining Potentially Predictive Biomarkers for Cystectomy-free Survival
Time Frame: as for outcome 7
Population: as for outcome 7
Arm/Group | 5-FU and Cisplatin + BID Irradiation | Gemcitabine + QD Irradiation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization to last follow-up. Maximum follow-up was 11.4 years.
Description: Adverse event population = eligible patients who started protocol treatment.
Groups:
- Arm I: Patients receive induction therapy comprising fluorouracil IV, cisplatin IV, and radiotherapy in weeks 1-4. Patients then undergo either radical cystectomy or receive consolidation therapy comprising fluorouracil IV, cisplatin IV, and radiotherapy in weeks 8-10.
- Arm II: Patients receive induction therapy comprising gemcitabine hydrochloride IV and radiotherapy in weeks 1-4. Patients then undergo either radical cystectomy or receive consolidation therapy comprising gemcitabine hydrochloride IV and radiotherapy in weeks 8-10.
Arm/Group | Arm I | Arm II
All-Cause Mortality (participants affected / at risk) | 16/33 | 11/33
Serious Adverse Events (participants affected / at risk) | 11/33 | 8/33
Other Adverse Events (participants affected / at risk) | 33/33 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=33) | Arm II (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Pain [other] (General disorders) | 1 | 0
Bladder infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1
Bladder infection [with unknown ANC] (Infections and infestations) | 1 | 0
Catheter related infection [with Grade 3-4 ANC] (Infections and infestations) | 0 | 1
Infection [other] (Infections and infestations) | 1 | 0
Pneumonia [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 1
Urinary tract infection [with unknown ANC] (Infections and infestations) | 1 | 0
Intraoperative complications (Injury, poisoning and procedural complications) | 1 | 0
Leukopenia (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=33) | Arm II (N=33)
Blood disorder (Blood and lymphatic system disorders) | 7 | 6
Hemoglobin decreased (Blood and lymphatic system disorders) | 28 | 30
Hemolysis (Blood and lymphatic system disorders) | 1 | 2
Cardiac disorder (Cardiac disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Eye disorder (Eye disorders) | 2 | 2
Vision blurred (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 11
Constipation (Gastrointestinal disorders) | 21 | 14
Diarrhea (Gastrointestinal disorders) | 23 | 28
Dry mouth (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 5 | 7
Flatulence (Gastrointestinal disorders) | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 6 | 11
Hemorrhoids (Gastrointestinal disorders) | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 26 | 24
Proctitis (Gastrointestinal disorders) | 1 | 5
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 2
Rectal pain (Gastrointestinal disorders) | 2 | 0
Stomach pain (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 12 | 7
Chest pain (General disorders) | 3 | 2
Chills (General disorders) | 1 | 6
Edema limbs (General disorders) | 6 | 4
Fatigue (General disorders) | 29 | 33
Fever (General disorders) | 4 | 10
General symptom (General disorders) | 3 | 1
Irritability (General disorders) | 0 | 2
Pain [other] (General disorders) | 13 | 8
Bladder infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 1 | 2
Bladder infection [with unknown ANC] (Infections and infestations) | 5 | 1
Urinary tract infection [with unknown ANC] (Infections and infestations) | 2 | 1
Intraoperative complications (Injury, poisoning and procedural complications) | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 7 | 18
Alkaline phosphatase increased (Investigations) | 10 | 8
Aspartate aminotransferase increased (Investigations) | 2 | 15
Creatinine increased (Investigations) | 14 | 7
Hyperbilirubinemia (Investigations) | 5 | 3
INR increased (Investigations) | 2 | 1
Laboratory test abnormal (Investigations) | 13 | 7
Leukopenia (Investigations) | 22 | 25
Lymphopenia (Investigations) | 19 | 14
Neutrophil count decreased (Investigations) | 19 | 16
Platelet count decreased (Investigations) | 20 | 20
Weight gain (Investigations) | 2 | 0
Weight loss (Investigations) | 8 | 7
Anorexia (Metabolism and nutrition disorders) | 12 | 16
Dehydration (Metabolism and nutrition disorders) | 11 | 10
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 25 | 17
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 13 | 8
Hypokalemia (Metabolism and nutrition disorders) | 10 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 17 | 13
Hyponatremia (Metabolism and nutrition disorders) | 19 | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 4
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Dizziness (Nervous system disorders) | 7 | 7
Headache (Nervous system disorders) | 7 | 9
Memory impairment (Nervous system disorders) | 2 | 0
Neurological disorder NOS (Nervous system disorders) | 5 | 3
Peripheral motor neuropathy (Nervous system disorders) | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 6
Taste alteration (Nervous system disorders) | 4 | 5
Agitation (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 4
Depression (Psychiatric disorders) | 7 | 3
Insomnia (Psychiatric disorders) | 17 | 9
Bladder pain (Renal and urinary disorders) | 2 | 2
Bladder spasm (Renal and urinary disorders) | 4 | 2
Cystitis (Renal and urinary disorders) | 6 | 12
Hemorrhage urinary tract (Renal and urinary disorders) | 5 | 3
Urethral pain (Renal and urinary disorders) | 1 | 3
Urinary frequency (Renal and urinary disorders) | 24 | 21
Urinary incontinence (Renal and urinary disorders) | 7 | 5
Urinary retention (Renal and urinary disorders) | 4 | 3
Urogenital disorder (Renal and urinary disorders) | 14 | 9
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 5
Pelvic pain (Reproductive system and breast disorders) | 1 | 2
Penile pain (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Hiccough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 4 | 3
Sweating (Skin and subcutaneous tissue disorders) | 0 | 2
Flushing (Vascular disorders) | 1 | 2
Hemorrhage (Vascular disorders) | 4 | 1
Hypertension (Vascular disorders) | 5 | 0
Hypotension (Vascular disorders) | 3 | 1
Phlebitis superficial (Vascular disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
Adverse event data was updated when outcome measure 5 was entered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-12-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT00777491/Prot_SAP_ICF_000.pdf